CLINICAL TRIAL: NCT01386944
Title: Non Interventional Observational Study to Collect Data for the Effect of Switching to Neupro® on Severity of Restless Leg Syndrome (RLS) Symptoms and Augmentation as Well as the Change in Treatment Regimen Used, in RLS Patients With Previous Augmentation
Brief Title: Effect on RLS Symptom Severity After Switching to Neupro® in Patients Who Previously Experienced Augmentation
Acronym: AURORA
Status: Completed | Type: Observational
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: SP1009
Record Dates: First submitted 2011-06-29; First posted 2011-07-01 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Restless Legs Syndrome
Keywords: Rotigotine; Neupro®; Augmentation; Restless Legs Syndrome; Moderate to severe; idiopathic; adults
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neupro® Treatment: Routine treatment (1,2,3 mg/24 h) as per approved label in the European Union (EU).

SUMMARY:
The objective is to assess the effect of Neupro® on the severity of Restless Leg Syndrome (RLS) symptoms and augmentation in patients with augmentation associated with previous oral dopaminergic therapy. In addition, the change in treatment regimen used when switching to Neupro® will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The adult patient has a diagnosis of moderate to severe idiopathic Restless Leg Syndrome (RLS)
* The patient must be experiencing augmentation due to a prior dopaminergic treatment
* The decision to prescribe Neupro® has been made by the physician independently of his/her decision to enroll the patient in the study
* Patient is informed and given ample time and opportunity to think about his/her participation in the study and has given written informed data consent

Exclusion Criteria:

* Patients diagnosed with secondary Restless Leg Syndrome (RLS) should not be enrolled in this observational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with a diagnosis of moderate to severe idiopathic Restless Leg Syndrome (RLS).
  Patient must be experiencing augmentation due to a prior dopaminergic treatment.
  Every consecutive, eligible patient to be treated with Neupro® as per physician's decision.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2011-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (18):
- Germany (18):
  - 12, Berlin
  - 4, Bremen
  - 18, Dresden
  - 20, Flensburg
  - 1, Kassel
  - 11, Marburg
  - 17, Marburg
  - 2, Mönchengladbach
  - 6, Münster
  - 7, Regensburg
  - 21, Remscheid
  - 15, Schriesheim
  - 10, Schwalmstadt
  - 3, Schwerin
  - 8, Tübingen
  - 16, Ulm
  - 9, Ulm
  - 19, Westerstede

REFERENCES:
- [Result] Trenkwalder C, Canelo M, Lang M, Schroeder H, Kelling D, Berkels R, Schollmayer E, Heidbrede T, Benes H. Management of augmentation of restless legs syndrome with rotigotine: a 1-year observational study. Sleep Med. 2017 Feb;30:257-265. doi: 10.1016/j.sleep.2015.10.006. Epub 2015 Nov 11. PMID 26896370

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This non-interventional study (NIS) was conducted in 18 specialized centres (medical practice and outpatient department) for neurology throughout Germany.
  The Participant Flow refers to the Enrolled Set (ES). The ES consists of all patients who provided informed consent.
Pre-assignment Details: The physician was to decide freely to treat the patient with Neupro®. In this context, the physician was not to change routine practice in reaching treatment decisions and in treating his/her patients because of the study. The observational period was 13 months per patient (adjustment period of medication switch plus 12 months of observation).
Period: Overall Study
Arm/Group | Neupro® Treatment
Started | 102
Completed | 46
Not Completed | 56
Not completed — Adverse Event | 26
Not completed — Lack of Efficacy | 14
Not completed — Lost to Follow-up | 8
Not completed — Unspecified reason | 8

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population refers to the Full Analysis Set (FAS). The FAS is a subset of the Safety Set and consists of all patients who received treatment with Neupro at least once and had a Visit 1 and at least one post-Visit 1 measurement on the primary variable documented.
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (11.1)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 31
Race/Ethnicity, Customized [Number; unit: participants]
  Scandinavian/Central European | 90
  Southern European | 5
  Missing | 2
Height [Mean (Standard Deviation); unit: centimeter] | 168.43 (9.48)
Weight [Mean (Standard Deviation); unit: kilogram] | 81.69 (15.93)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Visit 1) in Clinical Global Impression (CGI) (Item 1 - Severity of Illness) to Visit 2
Description: The CGI scales document a global assessment of the severity of RLS at single visits according to the treating physician. To this end the physician judges severity of disease by following a simple seven step severity rating scale:
  1. = Normal, not ill at all
  2. = Borderline ill
  3. = Mildly ill
  4. = Moderately ill
  5. = Markedly ill
  6. = Severely ill
  7. = Among the most extremely ill subjects
  A negative change from Baseline to Visit 2 indicates an improvement in CGI Item 1.
Time Frame: From Baseline up to 7 days
Population: The Analysis Population refers to the Full Analysis Set (FAS). The FAS is a subset of the Safety Set and consists of all patients who received treatment with Neupro at least once and had a Visit 1 and at least one post-Visit 1 measurement on the primary variable documented.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 89
score on a scale | -0.8 (1.1) [-1.0 to -0.5]
Statistical Analysis 1: Comparison: Neupro® Treatment; Test type: Superiority or Other; Hodges-Lehmann Estimate = -0.5, 95% CI 2-sided [-1.0 to -0.5]

2. Primary Outcome: Change From Baseline (Visit 1) in Clinical Global Impression (CGI) (Item 1 - Severity of Illness) to Visit 3
Description: The CGI scales document a global assessment of the severity of RLS at single visits according to the treating physician. To this end the physician judges severity of disease by following a simple seven step severity rating scale:
  1. = Normal, not ill at all
  2. = Borderline ill
  3. = Mildly ill
  4. = Moderately ill
  5. = Markedly ill
  6. = Severely ill
  7. = Among the most extremely ill subjects
  A negative change from Baseline to Visit 3 indicates an improvement in CGI Item 1.
Time Frame: From Baseline up to 28 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 77
score on a scale | -1.4 (1.3) [-1.5 to -1.0]
Statistical Analysis 1: Comparison: Neupro® Treatment; Test type: Superiority or Other; Hodges-Lehmann Estimate = -1.5, 95% CI 2-sided [-1.5 to -1.0]

3. Primary Outcome: Change From Baseline (Visit 1) in Clinical Global Impression (CGI) (Item 1 - Severity of Illness) to Visit 4
Description: The CGI scales document a global assessment of the severity of RLS at single visits according to the treating physician. To this end the physician judges severity of disease by following a simple seven step severity rating scale:
  1. = Normal, not ill at all
  2. = Borderline ill
  3. = Mildly ill
  4. = Moderately ill
  5. = Markedly ill
  6. = Severely ill
  7. = Among the most extremely ill subjects
  A negative change from Baseline to Visit 4 indicates an improvement in CGI Item 1.
Time Frame: From Baseline up to 4 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 58
score on a scale | -1.8 (1.2) [-2.0 to -1.5]
Statistical Analysis 1: Comparison: Neupro® Treatment; Test type: Superiority or Other; Hodges-Lehmann Estimate = -2.0, 95% CI [-2.0 to -1.5]

4. Primary Outcome: Change From Baseline (Visit 1) in Clinical Global Impression (CGI) (Item 1 - Severity of Illness) to Visit 5
Description: as for outcome 1
Time Frame: From Baseline up to 7 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 52
score on a scale | -2.0 (1.4) [-2.5 to -1.5]
Statistical Analysis 1: Comparison: Neupro® Treatment; Test type: Superiority or Other; Hodges-Lehmann Estimate = -2.0, 95% CI [-2.5 to -1.5]

5. Primary Outcome: Change From Baseline (Visit 1) in Clinical Global Impression (CGI) (Item 1 - Severity of Illness) to Visit 6
Description: The CGI scales document a global assessment of the severity of RLS at single visits according to the treating physician. To this end the physician judges severity of disease by following a simple seven step severity rating scale:
  1. = Normal, not ill at all
  2. = Borderline ill
  3. = Mildly ill
  4. = Moderately ill
  5. = Markedly ill
  6. = Severely ill
  7. = Among the most extremely ill subjects
  A negative change from Baseline to Visit 6 indicates an improvement in CGI Item 1.
Time Frame: From Baseline up to 10 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 45
score on a scale | -2.0 (1.3) [-2.5 to -1.5]
Statistical Analysis 1: Comparison: Neupro® Treatment; Test type: Superiority or Other; Hodges-Lehmann Estimate = -2.0, 95% CI [-2.5 to -1.5]

6. Primary Outcome: Change From Baseline (Visit 1) in Clinical Global Impression (CGI) (Item 1 - Severity of Illness) to Visit 7
Description: The CGI scales document a global assessment of the severity of RLS at single visits according to the treating physician. To this end the physician judges severity of disease by following a simple seven step severity rating scale:
  1. = Normal, not ill at all
  2. = Borderline ill
  3. = Mildly ill
  4. = Moderately ill
  5. = Markedly ill
  6. = Severely ill
  7. = Among the most extremely ill subjects
  A negative change from Baseline to Visit 7 indicates an improvement in CGI Item 1.
Time Frame: From Baseline up to 13 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 46
score on a scale | -1.8 (1.3) [-2.0 to -1.5]
Statistical Analysis 1: Comparison: Neupro® Treatment; Test type: Superiority or Other; Hodges-Lehmann Estimate = -2.0, 95% CI [-2.0 to -1.5]

7. Secondary Outcome: Change in Treatment Regimen Used for Switching to Neupro® up to 28 Days After Entering in the Study
Description: Case reports from clinical practice refer to different switching regimens for patients taking oral dopaminergics who experienced augmentation and then switched to Neupro®. The previous dopaminergic treatment might have been partly or completely down-titrated prior to switching to Neupro®. Physicians were requested to document the change of treatment at each recommended visit in the electronic Case Report Form (eCRF) considering their total clinical experience with this particular Restless Legs Syndrome (RLS) patients population. Documentation comprised changes in the RLS medication last prescribed, and the dosage of Neupro® and concomitant medications. The change of treatment regimen was entirely at the physicians' discretion.
Time Frame: From Baseline up to 28 days
Population: The Analysis Population refers to the Eligibility Completer Set (ECS). The ECS is a subset of the Completer Set excluding patients with Parkinson's disease and/or treated Polyneuropathy as concomitant disease identified by the preferred term (PT) of the MedDRA coding and patients treated with Neupro up to 4 weeks before Visit 1.
Measure: Number; unit: participants
Arm/Group | Neupro® Treatment
Number analyzed (Participants) | 43
participants
  Switch after "Drug holiday" | 5
  Overnight Switch | 23
  Overlapping Switch | 9
  No Switch | 6

ADVERSE EVENTS:
Time Frame: Adverse Events were reported from Day 1 up to 13 months.
Description: The Analysis Population refers to the Safety Set (SS). The Safety Set (SS) consists of all patients who have signed the consent form and who received treatment with Neupro at least once. Every Adverse Event occurring during the conduct of the study had to be entered in the respective electronic AE/SAE documentation form irrespective of causality.
Arm/Group | Neupro® Treatment
Serious Adverse Events (participants affected / at risk) | 9/99
Other Adverse Events (participants affected / at risk) | 40/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neupro® Treatment (N=99)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Acquired oesophageal web (Gastrointestinal disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Personality change (Psychiatric disorders) | 1 (1)
Acute stress disorder (Psychiatric disorders) | 1 (1)
Thinking abnormal (Psychiatric disorders) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thyroidectomy (Surgical and medical procedures) | 1 (1)
Arterial thrombosis limb (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neupro® Treatment (N=99)
Nausea (Gastrointestinal disorders) | 13 (15)
Application site erythema (General disorders) | 15 (17)
Application site reaction (General disorders) | 9 (9)
Application site pruritus (General disorders) | 8 (8)
Fatigue (General disorders) | 9 (9)
Headache (Nervous system disorders) | 6 (6)
Depression (Psychiatric disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days